CLINICAL TRIAL: NCT05086757
Title: Evaluation of Trauma Center-Based, Technology Enhanced Stepped Care Intervention for Adolescent Traumatic Injury Survivors.
Brief Title: Evaluation of Trauma Center-Based Intervention for Adolescent Traumatic Injury Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Children's of Alabama (Other); Boston Children's Hospital (Other); Prisma Health-Upstate (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111879; 1R01HD102336-01A1 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-10-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Injury; Technology; Posttraumatic Stress Disorder; Adolescents
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Trained interviewers blinded to condition will administer the 3-, 6-, and 12-month post-baseline assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma Resilience and Recovery Program (TRRP) (Experimental): Enrollment in TRRP which includes 3 major steps: (1) in-hospital education, brief risk reduction session, and tracking patients' emotional recovery via an automated text-messaging system, (2) conducting a 30-day screen via telephone to identify patients who are good candidates for psychological treatment, and (3) providing referral to formal mental health services, if needed.
  Interventions: Behavioral: TRRP
- Enhanced Usual Care (Active Comparator): Receive brief education about mental health after traumatic injury, educational materials about mental health recovery, and local referral information to assist treatment-seeking patients in seeking care
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: TRRP — Receive TRRP services
  Arms: Trauma Resilience and Recovery Program (TRRP)
Behavioral: Enhanced Usual Care — Participants will receive an educational flyer with service referrals
  Arms: Enhanced Usual Care

SUMMARY:
Pediatric traumatic injury (i.e., injury of sudden onset and severity requiring immediate attention) is the leading cause of death and morbidity among US adolescents and are associated with mental health and health risk outcomes, including posttraumatic stress and depression (affecting between 19-42%), deficits in physical recovery, social functioning and quality of life, which if unaddressed, may contribute to increased use of health care services. The investigators partnered with three accredited Level I and II pediatric trauma centers to conduct a multi-site hybrid 1 effectiveness-implementation trial with 300 adolescent (ages 12-17) traumatic injury patients to assess the extent to which the Trauma Resilience and Recovery Program (TRRP), a scalable and sustainable, technology-enhanced, multidisciplinary stepped model of care, promotes improvement in quality of life and emotional recovery and gather preliminary data on the potential for TRRP to be implemented in other Level I trauma centers. Directly in line with NICHD's Pediatric Trauma and Critical Illness Research and Training (PTCIB) Strategic Research and Training agenda, this study will provide valuable data on the efficacy, preliminary effectiveness and potential for implementation of an innovative, cost-effective, sustainable technology-enhanced intervention designed to address the unique needs of adolescent injury patients and mitigate short- and long-term impact of injury on mental health, quality of life, and overall well-being.

DETAILED DESCRIPTION:
Pediatric traumatic injury (i.e., injury of sudden onset and severity requiring immediate attention) is the leading cause of death and morbidity among US adolescents and are associated with mental health and health risk outcomes. Pediatric traumatic injuries are associated with medical and societal costs of $87 billion and elevates risk for a wide range of health risk consequences that affect quality of life, physical recovery, social functioning, and return to previous activities. The prevalence of PTSD and depression is high among pediatric traumatic injury patients; however, most pediatric trauma centers don't have the resources to implement models of care that address mental health following injury. Current guidelines by the American College of Surgeons (ACS) Committee on Trauma strongly recommend screening and addressing emotional recovery in traumatic injury patients. The ACS Committee on Trauma has identified this as a priority and likely will begin to mandate mental health programs in Level I and II pediatric trauma centers nationally. It is therefore critical that policy and practice is guided by the implementation and evaluation of scalable and sustainable models of care. In 2015 the investigators launched the Trauma Resilience and Recovery Program (TRRP), a scalable and sustainable, technology-enhanced, multidisciplinary stepped model of care - one of the few in the US - that provides early intervention and direct services to improve access to evidence-based mental health care after traumatic injury for children, adults and families. This model of care has been found to be feasible and acceptable to adolescent patients (ages 12-17) at each level of service. TRRP includes 3 major steps: (1) in-hospital education, brief risk reduction session, and tracking patients' emotional recovery via an automated text-messaging system, (2) conducting a 30-day screen via telephone to identify patients who are good candidates for psychological treatment, and (3) providing referral to best-practice telehealth-based or in-person assessment and treatment. The investigators partnered with three accredited Level I and II pediatric trauma centers and propose a multi-site hybrid 1 effectiveness-implementation trial with 300 adolescent (ages 12-17) traumatic injury patients to: 1) assess the extent to which TRRP promotes improvement in quality of life and emotional recovery and 2) gather preliminary data on the potential for TRRP to be implemented in other Level I trauma centers. Directly in line with NICHD's Pediatric Trauma and Critical Illness Research and Training (PTCIB) Strategic Research and Training agenda, this study will provide valuable data on the efficacy, preliminary effectiveness and potential for implementation of an innovative, cost-effective, sustainable technology-enhanced intervention designed to address the unique needs of adolescent injury patients and mitigate short- and long-term impact of injury on mental health, quality of life, and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* adolescent ages 12-17 admitted following traumatic injury
* scored significantly on the peritraumatic distress scale (PDI / ITSS)

Exclusion Criteria:

* if the injury was self-inflicted
* injuries are so severe, they prevent participation (e.g., head or spinal cord injuries that prevent verbal communication)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
The Child PTSD Symptom Scale, Caregiver/Child Version (CPSS) | 3 months post-baseline assessment
  The CPSS is a 26-item measure to assess PTSD diagnostic criteria and severity in youth. Responses are assessed using a 4-point Likert scale and a cutoff score of 31 can be used for identifying a probable PTSD diagnosis in children.
The Center for Epidemiological Studies Depression Scale (CES-DC) | 3 months post-baseline assessment
  This is a 20-item measure of depression with strong psychometric properties. Responses are assessed using a 4-point Likert scale and a cutoff score of 15 is suggestive of depressive symptoms in children and adolescents.

SECONDARY OUTCOMES:
Kessler 6 | Baseline, 3, 6, and 12-month post-baseline assessment
  This is a 6-item well-validated screening scale for nonspecific distress that demonstrates solid psychometric properties. Responses are assessed on a 5-point Likert scale and scores 13 or higher are suggestive of severe mental illness.
Peritraumatic Distress Inventory (PDI) | Baseline
  This is a 13-item measure with strong psychometric properties used to assess distress at the time of injury. Responses are on a 4-point Likert scale and scores above 15 are suggestive of peritraumatic distress. This measure has been validated with child traumatic injury survivors.
Injured Trauma Survivor Screen (ITSS) | Baseline
  This is a 9-item measure used to assess risk for development of posttraumatic stress symptoms following injury. Responses are in Yes/No format and a score of 2 on the PTSD questions suggest higher risk of developing PTSD and a score of 2 or more on the depression questions indicate higher risk for development of depression.
The Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) | Baseline, 3, 6, and 12-month post-baseline assessment
  This is a 3-item validated screen that identifies hazardous drinkers. The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Social Support Questionnaire, Short Form (SSQ6) | Baseline, 3, 6, and 12-month post-baseline assessment
  This is a 6-item measure of social support that includes both availability and satisfaction with social support.
Pediatric Quality of Life Inventory, Short Form (Peds QL-SF15) | Baseline, 3, 6, and 12-month post-baseline assessment
  This is a 15-item measure to assess health related QoL in youth with acute/chronic health conditions. Responses are assessed using a 5-point Likert scale with higher scores being indicative of higher health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Davidson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States